CLINICAL TRIAL: NCT00973323
Title: BAY 59-7939 (Factor Xa Inhibitor) Phase II Low Dose Study in Patients With Atrial Fibrillation
Brief Title: BAY59-7939 Japanese in Atrial Fibrillation (2nd)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12024
Record Dates: First submitted 2009-09-07; First posted 2009-09-09 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Atrial Fibrillation
Keywords: BAY59-7939; Rivaroxaban; Non-valvular atrial fibrillation; Japanese Patients; Phase II
MeSH Terms: conditions — Atrial Fibrillation | interventions — Rivaroxaban; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (Experimental)
  Interventions: Drug: Xarelto (Rivaroxaban, BAY59-7939)
- Arm 2 (Experimental)
  Interventions: Drug: Xarelto (Rivaroxaban, BAY59-7939)
- Arm 3 (Experimental)
  Interventions: Drug: Xarelto (Rivaroxaban, BAY59-7939)
- Arm 4 (Active Comparator)
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Xarelto (Rivaroxaban, BAY59-7939) — 2.5mg bid
  Arms: Arm 1
Drug: Xarelto (Rivaroxaban, BAY59-7939) — 5mg bid
  Arms: Arm 2
Drug: Xarelto (Rivaroxaban, BAY59-7939) — 10mg bid
  Arms: Arm 3
Drug: Warfarin — Dose-adjusted warfarin based on target INR values
  Arms: Arm 4

SUMMARY:
This study was a randomized, parallel group, open label trial using warfarin as comparator. Pharmacokinetics (PK) and pharmacodynamics (PD) were investigated only in BAY59-7939 groups (originally described in Japanese).

ELIGIBILITY:
Inclusion Criteria:

* Japanese subjects with non-valvular AF who met all of the following criteria:

  * Persistent or paroxysmal non-valvular AF with >/=2 episodes before enrollment, at least 1 of which had been verified by ECG recording within 4 weeks before randomization
  * Male subjects aged 20 years or older and postmenopausal female subjects
  * Subjects with at least one risk factor for thromboembolism or aged 60 years or older (Risk factor for thromboembolism: hypertension, diabetes mellitus, coronary artery disease, congestive heart failure).

Exclusion Criteria:

* History or presence of stroke or transient ischemic attack.
* History of intracerebral hemorrhage.
* History or presence of bleeding at randomization; intraocular or gastrointestinal bleeding within the last 6 months prior to randomization.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2005-09; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
(Safety) Incidence of bleeding | Throughout treatment and followup period
(PK/PD) BAY 59-7939 concentrations / Factor Xa activity, PT, PT-INR, PTT and HEPTEST | Day 14 and Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (10):
- Japan (10):
  - Fukui-shi, Fukui
  - Kurume, Fukuoka
  - Maebaru-chūō, Fukuoka
  - Kitahiroshima, Hokkaido
  - Kushiro, Hokkaido
  - Sapporo, Hokkaido
  - Nomi, Ishikawa-ken
  - Yokohama, Kanagawa
  - Ōita, Oita Prefecture
  - Tokorozawa, Saitama